CLINICAL TRIAL: NCT03194932
Title: A Phase I and Expansion Cohort Study of Venetoclax in Combination With Chemotherapy in Pediatric Patients With Refractory or Relapsed Acute Myeloid Leukemia
Brief Title: Study of Venetoclax in Combination With Chemotherapy in Pediatric Patients With Refractory or Relapsed Acute Myeloid Leukemia or Acute Leukemia of Ambiguous Lineage
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Gateway for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VENAML; NCI-2017-01129 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2017-06-19; First posted 2017-06-21 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; Cytarabine; Idarubicin; Methotrexate; Azacitidine

STUDY DESIGN:
Intervention Model Description: Participants receive venetoclax plus cytarabine alone or combination chemotherapy of cytarabine plus idarubicin.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): In Part 1, venetoclax with cytarabine will initially be given at dose level 1 and escalated based on tolerability. Idarubicin will be given only at dose level 4.
  Note: Part 1 has been completed.
  Two expansion cohorts will be enrolled:
  * Cohort A will be a group of 12 participants receiving the recommended phase 2 doses (RP2D) of venetoclax plus cytarabine.
  * Cohort B will be a group of 12 participants receiving the RP2D of venetoclax plus cytarabine and idarubicin.
  Intrathecal Triple Therapy (ITMHA) will be given prior to cycle 1. Patients without evidence of central nervous system (CNS) leukemia will receive no further IT therapy during cycle 1. Patients with CNS disease will receive weekly ITMHA beginning on day 8 until the cerebrospinal fluid becomes free of leukemia.
  Cohort C: Participants will receive venetoclax PO on days 1-21, azacitidine IV on days 1-7, and cytarabine Q12H on days 8-11.
  Interventions: Drug: Venetoclax; Drug: Cytarabine; Drug: Idarubicin; Drug: Intrathecal Triple Therapy; Drug: Azacitidine

INTERVENTIONS:
Drug: Venetoclax — Venetoclax will be given as oral tablets, which are intended to be swallowed intact and may not to be crushed or otherwise altered for administration, or as an oral suspension for patients who cannot swallow tablets.
  Other Names: Venclextra®; ABT-199
Drug: Cytarabine — Given intravenously (IV) or intrathecally (IT).
  Other Names: Cytosine arabinoside; Ara-C; Cytosar®
Drug: Idarubicin — Given IV.
  Other Names: Idamycin PFS
Drug: Intrathecal Triple Therapy — Given IT.
  Other Names: ITMHA; methotrexate/hydrocortisone/cytarabine
Drug: Azacitidine — Given IV.
  Other Names: VIDAZA®

SUMMARY:
The purpose of this study is to test the safety and determine the best dose of venetoclax and cytarabine when given with or without idarubicin in treating pediatric patients with acute myeloid leukemia (AML) that did not respond to treatment (refractory) or has come back after treatment (relapsed).

PRIMARY OBJECTIVE: Determine a tolerable combination of venetoclax plus chemotherapy in pediatric patients with relapsed or refractory AML or acute leukemia of ambiguous lineage. The primary endpoints are the recommended phase 2 doses (RP2D) of venetoclax plus cytarabine and venetoclax plus cytarabine and idarubicin.

SECONDARY OBJECTIVE: Estimate the overall response rate to the combination of venetoclax and chemotherapy in pediatric patients with relapsed or refractor AML or acute leukemia of ambiguous lineage. The secondary endpoints are the rates of complete remission (CR) and complete remission with incomplete count recovery (CRi) for patients treated at the RP2D.

DETAILED DESCRIPTION:
This study will be done in two parts:

* Part 1 - Dose Escalation: The goal of Part 1 of the study is to find the highest tolerable combination and recommended phase 2 doses (RP2D) of venetoclax plus cytarabine and venetoclax plus cytarabine and idarubicin that can be given to patients with leukemia.
* Part 2 - Dose Expansion: After determination of doses in Part 1, patients will be enrolled on Part 2 to look at the effects of venetoclax plus cytarabine and venetoclax plus cytarabine and idarubicin.

Depending on when participants enroll on the study, Part 1 participants will receive one of the following courses of therapy:

* Venetoclax daily on days 1-28; cytarabine every 12 hours on days 8-17; OR
* Venetoclax daily on days 1-28; cytarabine every 12 hours on days 8-11; OR
* Venetoclax daily on days 1-28; cytarabine every 12 hours on days 8-11; idarubicin once on day 8; OR
* Venetoclax daily on days 1-28; cytarabine every 12 hours on days 8-17; idarubicin once on day 8.

Part 2 participants will receive one of the following courses of therapy:

* Venetoclax daily on days 1-28; cytarabine - to be determined from Part 1 of the study; OR
* Venetoclax daily on days 1-28; cytarabine - to be determined from Part 1 of the study; idarubicin once on day 8.

The cytarabine dosage will be that found in Part 1 to be the highest safest dose.

Those participants receiving idarubicin will also receive dexrazoxane.

Note: Part 1 has been completed. Part 2 participants receive the following determined from Part 1 of the study:

* Venetoclax daily on days 1-28; cytarabine every 12 hours days 8-11 OR
* Venetoclax daily on days 1-28; cytarabine every 12 hours days 8-11; idarubicin once on day 8.

All participants on both Part 1 and Part 2 receive one intrathecal (IT) chemotherapy before starting the first cycle. Patients with CNS disease will receive weekly IT therapy until the cerebrospinal fluid becomes free of leukemia (minimum of 4 doses). Bone marrow aspiration and biopsy to assess response will be performed between days 28 and 42 of cycle 1. Patients who achieve complete remission/complete remission with incomplete count recovery/partial remission (CR/CRi/PR) and who do not experience unacceptable toxicity during cycle 1 may receive up to four cycles of chemotherapy.

Cohort C (Amendment 5.0): Treatment of participants enrolled in cohort C will include: Venetoclax daily on days 1-21; cytarabine every 12 hours days 8-11; azacytidine days 1-7. Participants will receive one intrathecal (IT) chemotherapy before starting the first cycle. Participants with CNS disease will receive weekly ITMHA until the cerebrospinal fluid becomes free of leukemia.

The rolling-6 design will be used to determine the safety of cohort C. After cohort C is deemed to be safe, additional patients will be enrolled, if necessary, so that at least 6 patients are treated in cohort C to confirm tolerability. After tolerability is confirmed, 6 additional patients will be treated to explore activity.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a diagnosis of AML or acute leukemia of ambiguous lineage (acute undifferentiated leukemia or mixed phenotype acute leukemia) and have refractory leukemia, defined as persistent leukemia after at least two courses of induction chemotherapy; or relapsed leukemia, defined as the re-appearance of leukemia after the achievement of remission.
* Patients in all categories above must have ≥ 5% blasts in the bone marrow as assessed by morphology or ≥ 1 blasts in the bone marrow as assessed by flow cytometry. However, if an adequate bone marrow sample cannot be obtained, patients may be enrolled if there is unequivocal evidence of leukemia with ≥ 5% blasts in the peripheral blood. In addition, patients in all categories must not be eligible to undergo curative therapy, such as immediate SCT, because of disease burden, time needed to identify a stem cell donor, or other reasons.

  * Adequate organ function defined as the following:
* Direct bilirubin ≤ 1.5 x institutional upper limit of normal (ULN)
* AST (SGOT) and ALT (SGPT) ≤ 4 x ULN
* Normal creatinine for age or a calculated creatinine clearance ≥ 60 mL/min/1.73 m2
* Left ventricular ejection fraction ≥ 40% or shortening fraction ≥ 25%

  * St. Jude patients must be between 2 years and ≤ 21 years of age, on therapy (active patient), or within 3 years of completion of therapy. Patients treated at collaborating sites must be ≤ 24 years old.
  * Performance status: Lansky ≥ 50 for patients who are ≤ 16 years old and Karnofsky ≥ 50% for patients who are > 16 years old.
  * Patients must have fully recovered from the acute effects of all prior therapy and cannot have evidence of graft-versus-host disease (GVHD)

Exclusion Criteria:

* Must not be pregnant or breastfeeding. Male or female of reproductive potential must agree to use effective contraception for the duration of study participation.
* Patients with Down syndrome, acute promyelocytic leukemia, juvenile myelomonocytic leukemia, or bone marrow failure syndromes are not eligible.
* Uncontrolled infection. Infections controlled on concurrent anti-microbial agents are acceptable, and anti-microbial prophylaxis per institutional guidelines are acceptable.
* Impairment of GI function or GI disease that may significantly alter the absorption of venetoclax.

Ages: 2 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 62 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2020-10-27 (Actual); Study Completion 2022-06-22 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated combination (MTC) | 28 days after start of therapy
  The MTC will be the highest intensity level at which six participants have been treated, with at most one participant experiencing an intensity-limiting toxicity.

SECONDARY OUTCOMES:
Complete Remission (CR) | Up to 6 weeks
  Will be assessed for the patients enrolled at the MTC (RP2D). Will be presented as a point estimate with a 95% exact binomial confidence interval.
Complete remission with incomplete count recovery (CRi) | Up to 6 weeks
  Will be assessed for the patients enrolled at the MTC (RP2D). Will be presented as a point estimate with a 95% exact binomial confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey E. Rubnitz, MD, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (3):
- United States (3):
  - Lucille Packard Children's Hospital Stanford University, Palo Alto, California
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - St. Jude Children's Research Hospital, Memphis, Tennessee

REFERENCES:
- [Derived] Badawi M, Gopalakrishnan S, Engelhardt B, Palenski T, Karol SE, Rubnitz JE, Menon R, Salem AH. Dosing of Venetoclax in Pediatric Patients with Relapsed Acute Myeloid Leukemia: Analysis of Developmental Pharmacokinetics and Exposure-Response Relationships. Clin Ther. 2024 Oct;46(10):759-767. doi: 10.1016/j.clinthera.2024.09.008. Epub 2024 Oct 5. PMID 39368878
- [Derived] Karol SE, Alexander TB, Budhraja A, Pounds SB, Canavera K, Wang L, Wolf J, Klco JM, Mead PE, Das Gupta S, Kim SY, Salem AH, Palenski T, Lacayo NJ, Pui CH, Opferman JT, Rubnitz JE. Venetoclax in combination with cytarabine with or without idarubicin in children with relapsed or refractory acute myeloid leukaemia: a phase 1, dose-escalation study. Lancet Oncol. 2020 Apr;21(4):551-560. doi: 10.1016/S1470-2045(20)30060-7. Epub 2020 Mar 11. PMID 32171069
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org